CLINICAL TRIAL: NCT00876811
Title: Raspberries and Human Health: A Short-term Intervention Trial Investigating the Effect of Daily Red Raspberry Consumption on Fasting Oxidative Stress Biomarkers
Brief Title: Effect of Red Raspberry Consumption on Fasting Oxidative Stress Biomarkers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Dr AV Rao, PhD, Professor Emeritus, Department of Nutritional Sciences, Faculty of Medicine, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22069
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Oxidative Stress
Keywords: raspberry; fruit; antioxidants; polyphenols; oxidative stress; dietary intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- one-cup (Experimental)
  Interventions: Dietary Supplement: individually quick frozen red raspberries
- two-cups (Experimental)
  Interventions: Dietary Supplement: individually quick frozen red raspberries
- four-cups (Experimental)
  Interventions: Dietary Supplement: individually quick frozen red raspberries

INTERVENTIONS:
Dietary Supplement: individually quick frozen red raspberries — Consumption of one-cup frozen red raspberries daily for four weeks, followed by a four week period of non-treatment.
  Arms: one-cup
Dietary Supplement: individually quick frozen red raspberries — Consumption of one-cup frozen red raspberries for two weeks, then consumption of two-cups frozen red raspberries for an additional two weeks, followed by four weeks of non-treatment.
  Arms: two-cups
Dietary Supplement: individually quick frozen red raspberries — Consumption of one-cup frozen red raspberries for two weeks, then consumption of four-cups frozen red raspberries for an addition two weeks, followed by four weeks of non-treatment.
  Arms: four-cups

SUMMARY:
The purpose of this study is determine whether daily consumption of frozen red raspberries can improve the antioxidant capacity of the blood and reduce the effects of oxidative stress, dose-dependently, in a healthy adult population.

DETAILED DESCRIPTION:
Red raspberries are an excellent source of numerous polyphenolic antioxidants. The bioactivity of these compounds have been implicated in many biological pathways and may function to reduce the risk of numerous chronic diseases. We are conducting an intervention study with frozen red raspberries on a healthy adult population in order to determine if raspberry polyphenols are bioavailable and bioactive in vivo. Twenty-four subjects (12 male and 12 female) will be recruited to participate and consume one-cup frozen red raspberries daily for two weeks, they then will randomly be assigned to consume either one, two or four cups of raspberries for another two weeks, this will be followed by four weeks of non-treatment. Blood samples and 12-hour urine collections will be taken in order to measure the concentration of raspberry polyphenols in response to treatment dose. Dose-dependent treatment effects on blood biomarkers for antioxidant capacity, oxidative stress, inflammation and other chronic disease risk factors will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults

Exclusion Criteria:

* obese (>30kg/m2)
* high blood pressure (140/90mmHg)
* allergic to raspberries
* pregnant or lactating
* history of chronic disease
* currently taking medication

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
serum TBARS | end of week 1, 3, 5 and 9
  an indicator of MDA levels, and therefore, lipid peroxidation

SECONDARY OUTCOMES:
serum antioxidant capacity (AOC) | end of week 1, 3, 5 and 9
  measured using the TEAC-ABTS radical cation assay
serum thiols | end of week 1, 3, 5 and 9
  measured using the DTNB assay, as an indicator of antioxidant levels in protein fraction

CONTACTS AND LOCATIONS:
Overall Officials: A V Rao, PhD, Principal Investigator — Department of Nutritional Sciences, University of Toronto
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada